CLINICAL TRIAL: NCT05701748
Title: EEG to Monitor Propofol Anesthetic Depth in Infants and Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-019941
Record Dates: First submitted 2023-01-17; First posted 2023-01-27 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Electroencephalography Spectral Edge Frequency; Anesthetic Depth
MeSH Terms: interventions — Stimuli Responsive Polymers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EEG SEF95 values in response to stimuli (Experimental): EEG SEF95 values that correspond to the three stimuli being applied, separately enrolled and analyzed for the 3-12mo and 13-24 age groups.
  Interventions: Other: Stimuli

INTERVENTIONS:
Other: Stimuli — placement of oral pacifier, electrical stimulation, and laryngoscopy

SUMMARY:
The goal of this study is monitor anesthetic depth of children undergoing propofol anesthesia using electroencephalography (EEG). The main questions it aims to answer are:

1. EEG spectral edge frequency (SEF95) readings where 50% of patients do not respond to three stimuli.
2. The propofol blood concentration that corresponds to each of the three EEG SEF95 readings Participants will undergo EEG monitoring, stimuli (placement of oral pacifier, electrical stimulation, and laryngoscopy), and blood collection.

DETAILED DESCRIPTION:
Sevoflurane inhalation and propofol intravenous anesthesia are the mainstays of delivering general anesthesia in children. Propofol anesthesia in children is gaining popularity due to fewer respiratory complications, less post-operative nausea vomiting and emergence delirium, compared to sevoflurane. However, unlike sevoflurane, the pharmacodynamics of propofol is less studied in infants and toddlers, particularly the biomarker for propofol brain effect site concentration (Ce), indicative of anesthetic depth. The lack of a real-time biomarker often results in over- or under-dosing of propofol in clinical practice. The goal of this study is to utilize electroencephalography (EEG) as the biomarker of propofol effect site concentration and clinical anesthetic depth, thereby improving the safety and efficacy of propofol anesthesia in this population. In infants and toddlers receiving propofol anesthesia, EEG will be recorded while the patient undergoes three stimuli used to assess anesthetic depth (placement of oral pacifier, electrical stimulation, and laryngoscopy). The EEG index (spectral edge frequency-SEF95) where 50% of patients (ED50) do not respond to each of the three stimuli will be determined as the biomarker of propofol clinical anesthetic depth. In the same cohort, the regression between EEG SEF95 and plasma propofol levels will be determined to assess relationship between EEG SEF95 and propofol Ce.

ELIGIBILITY:
Inclusion Criteria:

1. Children 3 to 24 month old undergoing surgery.
2. Planned laryngoscopy and endotracheal intubation or laryngeal mask airway (LMA) placement for clinical care.
3. Planned propofol anesthesia for anesthesia maintenance.
4. American Society of Anesthesiologists (ASA ) < III.
5. Muscle relaxant not indicated per planned clinical care for laryngoscopy/intubation or LMA.
6. Anticipated surgery duration approximately < 2h40min

Exclusion Criteria:

1. Patients undergoing emergency surgery.
2. Known severe neurological disease which might result in abnormal EEG SEF.
3. Deformities of forehead (difficult EEG sensor placement).
4. Known difficult airway.
5. Allergy to propofol.
6. Attending anesthesiologist on record caring for patient plans to administer additional IV medication besides propofol during study phase.
7. Currently on anti-seizure medication (might alter propofol pharmacodynamics).

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
EEG SEF95 value where 50% of infants do not respond to placement of oral pacifier | Once SEF95 stabilizes at oral pacifier target SEF95 +/- 1Hz for at least one minute
  Observation in OR and EEG data analysis
EEG SEF95 value where 50% of infants do not respond to electrical stimulation | Once SEF95 stabilizes at electrical stimulation target SEF95 +/- 1Hz for at least one minute
  Observation in OR and EEG data analysis
EEG SEF95 value where 50% of infants do not respond to laryngoscopy | Once SEF95 stabilizes at laryngoscopy target SEF95 +/- 1Hz for at least one minute
  Observation in OR and EEG data analysis

SECONDARY OUTCOMES:
Correlation of propofol blood concentration with EEG SEF95 | Once SEF95 stabilizes for at least one minute
  Blood collection and testing

CONTACTS AND LOCATIONS:
Overall Officials: Ian Yuan, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Brioni JD, Varughese S, Ahmed R, Bein B. A clinical review of inhalation anesthesia with sevoflurane: from early research to emerging topics. J Anesth. 2017 Oct;31(5):764-778. doi: 10.1007/s00540-017-2375-6. Epub 2017 Jun 5. PMID 28585095
- [Background] Chidambaran V, Costandi A, D'Mello A. Propofol: a review of its role in pediatric anesthesia and sedation. CNS Drugs. 2015 Jul;29(7):543-63. doi: 10.1007/s40263-015-0259-6. PMID 26290263
- [Background] Morse J, Hannam JA, Cortinez LI, Allegaert K, Anderson BJ. A manual propofol infusion regimen for neonates and infants. Paediatr Anaesth. 2019 Sep;29(9):907-914. doi: 10.1111/pan.13706. Epub 2019 Aug 12. PMID 31325395
- [Background] Sepulveda P, Cortinez LI, Saez C, Penna A, Solari S, Guerra I, Absalom AR. Performance evaluation of paediatric propofol pharmacokinetic models in healthy young children. Br J Anaesth. 2011 Oct;107(4):593-600. doi: 10.1093/bja/aer198. Epub 2011 Jul 9. PMID 21743068
- [Background] Oberer C, von Ungern-Sternberg BS, Frei FJ, Erb TO. Respiratory reflex responses of the larynx differ between sevoflurane and propofol in pediatric patients. Anesthesiology. 2005 Dec;103(6):1142-8. doi: 10.1097/00000542-200512000-00007. PMID 16306725
- [Background] Chandler JR, Myers D, Mehta D, Whyte E, Groberman MK, Montgomery CJ, Ansermino JM. Emergence delirium in children: a randomized trial to compare total intravenous anesthesia with propofol and remifentanil to inhalational sevoflurane anesthesia. Paediatr Anaesth. 2013 Apr;23(4):309-15. doi: 10.1111/pan.12090. PMID 23464658
- [Background] Sneyd JR, Carr A, Byrom WD, Bilski AJ. A meta-analysis of nausea and vomiting following maintenance of anaesthesia with propofol or inhalational agents. Eur J Anaesthesiol. 1998 Jul;15(4):433-45. doi: 10.1046/j.1365-2346.1998.00319.x. PMID 9699101
- [Background] Sarner JB, Levine M, Davis PJ, Lerman J, Cook DR, Motoyama EK. Clinical characteristics of sevoflurane in children. A comparison with halothane. Anesthesiology. 1995 Jan;82(1):38-46. doi: 10.1097/00000542-199501000-00006. PMID 7832332
- [Background] Lerman J, Sikich N, Kleinman S, Yentis S. The pharmacology of sevoflurane in infants and children. Anesthesiology. 1994 Apr;80(4):814-24. doi: 10.1097/00000542-199404000-00014. PMID 8024136
- [Background] Kim TK, Niklewski PJ, Martin JF, Obara S, Egan TD. Enhancing a sedation score to include truly noxious stimulation: the Extended Observer's Assessment of Alertness and Sedation (EOAA/S). Br J Anaesth. 2015 Oct;115(4):569-77. doi: 10.1093/bja/aev306. PMID 26385665
- [Background] Fuentes R, Cortinez I, Ibacache M, Concha M, Munoz H. Propofol concentration to induce general anesthesia in children aged 3-11 years with the Kataria effect-site model. Paediatr Anaesth. 2015 Jun;25(6):554-9. doi: 10.1111/pan.12657. Epub 2015 Apr 16. PMID 25880448
- [Background] Xu T, Kurth CD, Yuan I, Vutskits L, Zhu T. An approach to using pharmacokinetics and electroencephalography for propofol anesthesia for surgery in infants. Paediatr Anaesth. 2020 Dec;30(12):1299-1307. doi: 10.1111/pan.14021. Epub 2020 Oct 28. PMID 32965066
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Background] Chan MTV, Hedrick TL, Egan TD, Garcia PS, Koch S, Purdon PL, Ramsay MA, Miller TE, McEvoy MD, Gan TJ; Perioperative Quality Initiative (POQI) 6 Workgroup. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on the Role of Neuromonitoring in Perioperative Outcomes: Electroencephalography. Anesth Analg. 2020 May;130(5):1278-1291. doi: 10.1213/ANE.0000000000004502. PMID 31764163
- [Background] Yuan I, Xu T, Skowno J, Zhang B, Davidson A, von Ungern-Sternberg BS, Sommerfield D, Zhang J, Song X, Zhang M, Zhao P, Liu H, Jiang Y, Zuo Y, de Graaff JC, Vutskits L, Olbrecht VA, Szmuk P, Kurth CD; BRAIN Collaborative Investigators. Isoelectric Electroencephalography in Infants and Toddlers during Anesthesia for Surgery: An International Observational Study. Anesthesiology. 2022 Aug 1;137(2):187-200. doi: 10.1097/ALN.0000000000004262. PMID 35503999
- [Background] FDA. Propofol FDA https://www.accessdata.fda.gov/drugsatfda_docs/label/2014/019627s062lbl.pdf. Accessed
- [Background] Yuan I, Xu T, Kurth CD. Using Electroencephalography (EEG) to Guide Propofol and Sevoflurane Dosing in Pediatric Anesthesia. Anesthesiol Clin. 2020 Sep;38(3):709-725. doi: 10.1016/j.anclin.2020.06.007. PMID 32792193
- [Background] Hayashi K, Shigemi K, Sawa T. Neonatal electroencephalography shows low sensitivity to anesthesia. Neurosci Lett. 2012 May 31;517(2):87-91. doi: 10.1016/j.neulet.2012.04.028. Epub 2012 Apr 19. PMID 22542892
- [Background] Davidson AJ, Wong A, Knottenbelt G, Sheppard S, Donath S, Frawley G. MAC-awake of sevoflurane in children. Paediatr Anaesth. 2008 Aug;18(8):702-7. doi: 10.1111/j.1460-9592.2008.02664.x. PMID 18613929
- [Background] Zbinden AM, Maggiorini M, Petersen-Felix S, Lauber R, Thomson DA, Minder CE. Anesthetic depth defined using multiple noxious stimuli during isoflurane/oxygen anesthesia. I. Motor reactions. Anesthesiology. 1994 Feb;80(2):253-60. doi: 10.1097/00000542-199402000-00004. PMID 8311307
- [Background] Inomata S, Kihara S, Yaguchi Y, Baba Y, Kohda Y, Toyooka H. Reduction in standard MAC and MAC for intubation after clonidine premedication in children. Br J Anaesth. 2000 Nov;85(5):700-4. doi: 10.1093/bja/85.5.700. PMID 11094583
- [Background] Dixon W. The up-and-down method for small samples. Journal of the American Statistical Association. 1965;60(312):967-978.
- [Background] Pace NL, Stylianou MP. Advances in and limitations of up-and-down methodology: a precis of clinical use, study design, and dose estimation in anesthesia research. Anesthesiology. 2007 Jul;107(1):144-52. doi: 10.1097/01.anes.0000267514.42592.2a. PMID 17585226
- [Background] Gorges M, Zhou G, Brant R, Ansermino JM. Sequential allocation trial design in anesthesia: an introduction to methods, modeling, and clinical applications. Paediatr Anaesth. 2017 Mar;27(3):240-247. doi: 10.1111/pan.13088. Epub 2017 Feb 17. PMID 28211193
- [Background] Kataria BK, Ved SA, Nicodemus HF, Hoy GR, Lea D, Dubois MY, Mandema JW, Shafer SL. The pharmacokinetics of propofol in children using three different data analysis approaches. Anesthesiology. 1994 Jan;80(1):104-22. doi: 10.1097/00000542-199401000-00018. PMID 8291699
- [Background] Coppens MJ, Eleveld DJ, Proost JH, Marks LA, Van Bocxlaer JF, Vereecke H, Absalom AR, Struys MM. An evaluation of using population pharmacokinetic models to estimate pharmacodynamic parameters for propofol and bispectral index in children. Anesthesiology. 2011 Jul;115(1):83-93. doi: 10.1097/ALN.0b013e31821a8d80. PMID 21555936
- [Background] Absalom A, Amutike D, Lal A, White M, Kenny GN. Accuracy of the 'Paedfusor' in children undergoing cardiac surgery or catheterization. Br J Anaesth. 2003 Oct;91(4):507-13. doi: 10.1093/bja/aeg220. PMID 14504151
- [Background] Rigouzzo A, Girault L, Louvet N, Servin F, De-Smet T, Piat V, Seeman R, Murat I, Constant I. The relationship between bispectral index and propofol during target-controlled infusion anesthesia: a comparative study between children and young adults. Anesth Analg. 2008 Apr;106(4):1109-16, table of contents. doi: 10.1213/ane.0b013e318164f388. PMID 18349180
- [Background] Sahinovic MM, Struys MMRF, Absalom AR. Clinical Pharmacokinetics and Pharmacodynamics of Propofol. Clin Pharmacokinet. 2018 Dec;57(12):1539-1558. doi: 10.1007/s40262-018-0672-3. PMID 30019172
- [Background] Olbrecht VA, Jiang Y, Viola L, Walter CM, Liu H, Kurth CD. Characterization of the functional near-infrared spectroscopy response to nociception in a pediatric population. Paediatr Anaesth. 2018 Feb;28(2):103-111. doi: 10.1111/pan.13301. Epub 2017 Dec 27. PMID 29280254
- [Background] Hammer GB, Litalien C, Wellis V, Drover DR. Determination of the median effective concentration (EC50) of propofol during oesophagogastroduodenoscopy in children. Paediatr Anaesth. 2001;11(5):549-53. doi: 10.1046/j.1460-9592.2001.00731.x. PMID 11696118
- [Background] Yuan I, Landis WP, Topjian AA, Abend NS, Lang SS, Huh JW, Kirschen MP, Mensinger JL, Zhang B, Kurth CD. Prevalence of Isoelectric Electroencephalography Events in Infants and Young Children Undergoing General Anesthesia. Anesth Analg. 2020 Feb;130(2):462-471. doi: 10.1213/ANE.0000000000004221. PMID 31107263
- [Background] Disma N, Veyckemans F, Virag K, Hansen TG, Becke K, Harlet P, Vutskits L, Walker SM, de Graaff JC, Zielinska M, Simic D, Engelhardt T, Habre W; NECTARINE Group of the European Society of Anaesthesiology Clinical Trial Network; Austria; Belgium; Croatia; Czech Republic; Denmark; Estonia; Finland; France; Germany; Greece; Hungary; Ireland; Italy; Latvia; Lithuania; Luxembourg; Malta; Netherlands; Norway; Poland; Portugal; Romania; Serbia; Slovakia; Slovenia; Spain; Switzerland; Turkey; Ukraine; United Kingdom. Morbidity and mortality after anaesthesia in early life: results of the European prospective multicentre observational study, neonate and children audit of anaesthesia practice in Europe (NECTARINE). Br J Anaesth. 2021 Jun;126(6):1157-1172. doi: 10.1016/j.bja.2021.02.016. Epub 2021 Apr 1. PMID 33812668

DOCUMENTS (2):
  • Study Protocol (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT05701748/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT05701748/SAP_002.pdf